CLINICAL TRIAL: NCT05413499
Title: BRAINI2-Paediatric : Blood Biomarkers to Improve Management of Children With Traumatic Brain Injury: a European, Prospective, Multicentre Clinical Study
Brief Title: Blood Biomarkers to Improve Management of Children With Traumatic Brain Injury
Acronym: BRAINI2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC21_0595
Record Dates: First submitted 2022-06-01; First posted 2022-06-10 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Traumatic Brain Injury
Keywords: TBI / Biomarkers / paediatric
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Biomarkers research — For a part of the included population, the children with a mTBI and without indication of CT scan, a non-routine blood sample will be planned

SUMMARY:
Mild traumatic brain injury (TBI), defined by a Glasgow Coma Scale (GCS) score of 13 to 15, is the cause of many consultations in paediatric emergency departments (1), even though it is a rare cause of acute complication: approximately 10% of children present with intracranial lesions (ICL) on the CT scan and less than 1% require neurosurgical intervention (2). Although ICLs remain a serious complication requiring rapid diagnosis, brain CT scans, the gold standard diagnostic test, cannot be performed routinely because many children would be unnecessarily exposed to ionising radiation associated with an increased risk of cancer (3). In recent years, several clinical decision rules for the management of mTBI have therefore been developed with the aim of identifying children at high or very low risk of ICL in order to better target CT scan indications. Despite this, the rate of CT scans performed has remained high, up to 35%, and has not decreased with the application of these clinical decision rules (4).

Furthermore, even though the majority of children and adolescents recover quickly after mTBI, nearly 30% will present symptoms such as headaches, dizziness, asthenia, memory, concentration or sleep disorders persisting beyond one month with a possible impact on their quality of life (5). Thus, there is a need to develop new strategies to (i) limit the use of CT scans while minimising the risk of late diagnosis of ICL, (ii) identify children with a higher risk of adverse outcome and/or post-concussive symptoms.

One of the most promising strategies is the use of brain-based blood biomarkers. This study therefore aims to provide new knowledge on two of them, GFAP and UCH-L1 (6,7), in particular by using an automated test combining them (the VIDAS® TBI test developed by bioMérieux) in order to improve the management of CT in the paediatric population at the diagnostic and prognostic levels.

ELIGIBILITY:
Inclusion Criteria:

Children and adolescents <18 years old Consent from one of the parents of the child or from holder of parental responsibility Consent from the child or adolescent Parental affiliation with an appropriate health insurance system

1. TBI population

   * Admission within 24 hours of the injury
   * Ability to follow-up by telephone, mail or email
   * For the mTBI group:

     * GCS score of 13-15 on admission
     * Indication for cerebral CT scan according to national or local guidelines or the in-charge physician OR diagnosis of concussion consistent with the fourth Zurich consensus statement (9) . Concussion was defined as a complex pathophysiological process caused by a direct blow to the head, face, neck, or elsewhere on the body with an impulsive force transmitted to the head (which may or may not have involved loss of consciousness), resulting in a brain injury with one or more symptoms in one or more of the following clinical domains: somatic, cognitive, emotional or behavioural, or sleep. To objectively help diagnose concussion, the validated Acute Concussion Evaluation (ACE) questionnaire (10) for children with mTBI will be used, the presence of ≥ 1 symptom on the ACE defines concussion.
   * For the moderate or severe TBI group:

     * GCS score of 3-12 on admission
     * Indication for cerebral CT scan according to national or local guidelines or the in-charge physician
2. Non-TBI control paediatric population

   * Admission for any reason other than TBI
   * Indication of blood sampling for their routine management
   * GCS score of 15
   * Otherwise healthy, i.e. without chronic pathology

Exclusion Criteria:

1. TBI population

   * Time of injury unknown or exceeding 24 hours
   * Blood sampling not possible within 24 hours after the injury or 6 hours after the CT scan, if applicable
   * Penetrating brain injury with skull fracture
   * Pre-existing neurological disorders affecting the assessment of neurological outcome, seizure disorder/epilepsy, brain tumour, history of neurosurgery, stroke, encephalopathy
   * Venepuncture not feasible
   * Pregnant woman
   * Intoxication
   * No clear primary mechanism of trauma
   * No possibility for transferring CT scan images to the centralised platform in case of neuroimaging only performed in an outside hospital before transfer
   * Participation in another interventional research study
2. Non-TBI control paediatric population

   * Pre-existing neurological disorders, seizure disorder/epilepsy, brain tumour, history or indication of neurosurgery, stroke, encephalopathy
   * History of TBI
   * Orthopaedic trauma or surgery within the last month
   * Suspected meningitidis or encephalitis
   * Venepuncture not feasible
   * Pregnant woman
   * Intoxication
   * Participation in another interventional research study

Ages: 0 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2880 (Estimated)
Dates: Start 2022-08-02 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) of GFAP and UCHL-1 used separately and in combination to detect the presence or absence of ICL on CT scan | Day 0

SECONDARY OUTCOMES:
Prediction of early and mid-term prognosis after TBI : Number of participants with Early clinical worsening | 72 hours after TBI
  Early clinical worsening defined by the occurrence of death from TBI, neurosurgical intervention, intubation for TBI, or hospital admission of two nights or more associated with ICL on CT scan for persistent neurological symptoms such as persistent alteration in mental status, recurrent emesis due to TBI, persistent severe headache, or ongoing seizure management (8), within 72 hours after TBI.
Prediction of early and mid-term prognosis after TBI : Glasgow Outcome Scale-Extended, paediatric version (GOS-E Peds) | Month 1, Month 3
  Neurological outcome: Glasgow Outcome Scale-Extended, paediatric version (GOS-E Peds)
Prediction of early and mid-term prognosis after TBI : ost-concussion symptoms: Rivermead Post-Concussion Symptoms Questionnaire (RPQ) | Month 1, Month 3
  Post-concussion symptoms: Rivermead Post-Concussion Symptoms Questionnaire (RPQ)
Prediction of early and mid-term prognosis after TBI : Health related quality of life: PedsQL questionnaire | Month 1, Month 3
  Health related quality of life: PedsQL questionnaires
Prediction of early and mid-term prognosis after TBI : Serum GFAP and UCH-L1 concentrations | Day 0
  Comparison of serum GFAP and UCH-L1 concentrations according to the TBI severity groups, i.e. mild (GCS score of 13-15), moderate (GCS score of 9-12) or severe (GCS score of 3-8)
Establishment of age-appropriate physiological reference values | Day 0
  Measure of serum GFAP and UCH-L1 concentrations in three age groups (under 2 years old, 2-9 years old and aged 10 and over) in a non-TBI control paediatric population

CONTACTS AND LOCATIONS:
Overall Officials: Fleur LORTON, Principal Investigator — Nantes University Hospital
Locations (20):
- France (15):
  - Brest University Hospital, Brest
  - Clermont-Ferrand University Hospital, Clermont-Ferrand
  - Louis Mourier Hospital (AP-HP), Colombes
  - Grenoble University Hospital, Grenoble
  - La Roche/Yon Hospital, La Roche-sur-Yon
  - Lille University Hospital, Lille
  - Limoges University Hospital, Limoges
  - Lorient Hospital, Lorient
  - Montpellier University Hospital, Montpellier
  - Nantes University Hospital, Nantes
  - Armand Trousseau hospital (AP-HP), Paris
  - Robert Debré Hospital (AP-HP), Paris
  - Rennes University Hospital, Rennes
  - Saint Etienne University Hospital, Saint-Etienne
  - Saint Nazaire Hospital, Saint-Nazaire
- Klinikum rechts der Isar, Technical University of Munich, Munich, Germany
- Spain (3):
  - Hospital Universitari Vall d'Hebron (ICS), Barcelona
  - Hospital 12 de Octubre, Madrid
  - Hospital Infantil Universitario Nino Jesus, Madrid
- Luzerner Kantonsspital, Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lorton F, Lagares A, de la Cruz J, Mejan O, Pavlov V, Sapin V, Poca MA, Lehner M, Biberthaler P, Chauvire-Drouard A, Gras-Le-Guen C, Scherdel P; BRAINI-2 paediatric Collaborative group; Collaborators. Performance of glial fibrillary acidic protein (GFAP) and ubiquitin carboxy-terminal hydrolase L1 (UCH-L1) biomarkers in predicting CT scan results and neurological outcomes in children with traumatic brain injury (BRAINI-2 paediatric study): protocol of a European prospective multicentre study. BMJ Open. 2024 May 15;14(5):e083531. doi: 10.1136/bmjopen-2023-083531. PMID 38754888